CLINICAL TRIAL: NCT01982071
Title: A Multi-center, Open-label, Non-comparative Study to Evaluate the Efficacy and Safety of Micafungin Against Invasive Candidiasis or Candidemia (CFDA Commitment)
Brief Title: A Study to Evaluate the Efficacy and Safety of Micafungin Against Invasive Candidiasis or Candidemia
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to administrative reasons
Sponsor: Astellas Pharma China, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACN-MA-MYC-IC-2012
Record Dates: First submitted 2013-11-06; First posted 2013-11-13 (Estimated); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Candidemia; Candidiasis
Keywords: Micafungin; candidiasis; candidemia; Open-label design
MeSH Terms: conditions — Candidemia; Candidiasis | interventions — Micafungin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment group (Experimental): Intravenous (IV)
  Interventions: Drug: Micafungin

INTERVENTIONS:
Drug: Micafungin — Intravenous (IV)

SUMMARY:
To evaluate the efficacy and safety of intravenous micafungin for the treatment of patients with proven or probable fungal infections caused by Candida sp. (Fungemia, respiratory mycosis, gastrointestinal mycosis) in adult patients in China.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis criteria of probable candida infection: Risk factors + Clinical Manifestations + positive findings including microbiologic test
* The diagnosis criteria of proven candida infection: Risk factors + Clinical Manifestation + positive findings including microbiologic test + tissue culture or pathological examination results
* The following 3 criteria must be met is a patient is diagnosed as probable candida pneumonia:

  1. Risk factor (s) of infection
  2. Clinical manifestations of infection and the pulmonary infection cannot be explained by other pathogenic infections
  3. Two or more positive sputum culture for Candida

Exclusion Criteria:

* Patient received any other antifungal drug within 1 month prior to enrollment.
* HIV positive patient
* Patients with organ transplant
* Patients with agranulocytosis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2013-09-26 (Actual); Primary Completion 2015-08-28 (Actual); Study Completion 2015-08-28 (Actual)

PRIMARY OUTCOMES:
Overall success rate | up to 8 weeks
  success rate is calculated as (number of success patients/number of patients for efficacy evaluation × 100% at end of treatment)

SECONDARY OUTCOMES:
Safety assessed by the incidence of adverse events | up to 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Principal Investigator — Astellas Pharma Inc
Locations (15):
- China (15):
  - Beijing
  - Changsha
  - Chengdu
  - Fuzhou
  - Guangzhou
  - Harbin
  - Hengyang
  - Jinan
  - Nanjing
  - Shanghai
  - Shaoyang
  - Shenyang
  - Tianjin
  - Xi'an
  - Xiamen

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on Astellas Clinical Study Results website — https://www.astellasclinicalstudyresults.com/study.aspx?ID=172